CLINICAL TRIAL: NCT04908397
Title: Carnitine Consumption and Augmentation in Pulmonary Arterial Hypertension
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Anna Hemnes, Associate Professor of Allergy, Pulmonary, and Critical Care Medicine, Vanderbilt University Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 210899
Record Dates: First submitted 2021-05-17; First posted 2021-06-01 (Actual); Results first posted 2025-02-13 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Pulmonary Arterial Hypertension; Familial Primary Pulmonary Hypertension; Primary Pulmonary Hypertension; Lung Diseases; Carnitine Nutritional Deficiency
MeSH Terms: conditions — Pulmonary Arterial Hypertension; Familial Primary Pulmonary Hypertension; Lung Diseases | interventions — Carnitine

STUDY DESIGN:
Intervention Model Description: This is a single-center, prospective study enrolling 10 PAH patients. All eligible participants will be given carnitine supplements for 2 weeks.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Supplement (Experimental): Form: 500 mg L-carnitine tablet Dosage: Subjects 50-90kg: 3g/day Subjects <50kg or >90kg: 50mg/kg/day Frequency: twice a day for 2 weeks
  Interventions: Dietary Supplement: L-carnitine

INTERVENTIONS:
Dietary Supplement: L-carnitine — supplement provided twice a day for 2 weeks
  Other Names: Carnitine; Carnitor

SUMMARY:
In preparation for a future mechanistic study, investigators now propose to test the specific hypothesis that carnitine consumption is not reduced in PAH, that plasma carnitine levels are stable over time in PAH and that carnitine supplementation in PAH can increase plasma carnitine and thereby delivery of carnitine to the RV and possibly improve RV function. Investigators propose three aims in humans to test this mechanistic hypothesis, 1) Measure the oral consumption of carnitine in human PAH. This aim will use food diaries and carnitine supplement use questionnaires in PAH patients to test the hypothesis that carnitine supplementation is uncommon in PAH and food consumption is adequate. Aim 2) Measure the stability over time in plasma carnitine levels in PAH patients. This aim will test the hypothesis that plasma carnitine is not affected by disease severity and is stable over time in PAH patients. Investigators will measure plasma carnitine concentration and markers of fatty acid oxidation at Visit 1 and Visit 2. 3) Perform a mechanistic pilot study using carnitine supplementation to enhance circulating carnitine in PAH. This small pilot study will test the hypothesis that carnitine supplementation increases plasma carnitine (primary endpoint) and will test for physiologic effects using six minute walk testing, echocardiography and plasma markers of lipid metabolism.

DETAILED DESCRIPTION:
Right ventricular (RV) failure is the most common cause of death in pulmonary arterial hypertension (PAH). No RV-specific therapies are available, in part because the underlying mechanisms of RV failure are poorly understood. A growing body of evidence suggests that metabolic abnormalities may underlie RV dysfunction in PAH. Interventions against metabolic dysfunction in PAH may protect against RV failure. Investigators in the PH research group have identified abnormalities in fatty acid (FA) metabolism in PAH that overlap considerably with disorders of carnitine deficiency. Carnitine links to an acyl group, which is required to transport FAs across the mitochondrial membrane to undergo beta-oxidation, the predominate source of ATP production in the human heart. Inborn errors of carnitine metabolism and acquired carnitine deficiency are associated with cardiomyopathy. Acquired deficiency primarily occurs via binding of carnitine to excess circulating fatty acids or renal wasting. Carnitine deficiency and PAH are both associated with insulin resistance, myocardial lipotoxicity, and mitochondrial oxidative stress. Carnitine supplementation in humans and animal models of cardiometabolic dysfunction reverses these abnormalities but has not been studied in PAH. In published work, investigators found that in RV samples from humans with PAH, there is a marked (up to 300-fold) reduction in acylcarnitines along with increased long-chain fatty acids. Investigators also a found a two-fold increase in circulating fatty acids FAs in humans with PAH, indicating increased delivery to the myocardium. As a consequence of unchecked fatty acid accumulation, investigators observed 7-fold higher RV lipid content and markers of lipotoxicity. These observations suggest there is inadequate carnitine substrate to bind fatty acids and facilitate their transport across the mitochondrial membrane in the human PAH RV.

The investigator's overarching hypothesis is that in human PAH, RV function can be improved by augmenting carnitine substrate availability to improve outcomes. In preparation for a future mechanistic study, Vanderbilt PAH research investigators now propose to test the specific hypothesis that carnitine consumption is not reduced in PAH, that plasma carnitine levels are stable over time in PAH and that carnitine supplementation in PAH can increase plasma carnitine and thereby delivery of carnitine to the RV and possibly improve RV function. Investigators propose three aims in humans to test this mechanistic hypothesis, 1) Measure the oral consumption of carnitine in human PAH. This aim will use food diaries and carnitine supplement use questionnaires in PAH patients to test the hypothesis that carnitine supplementation is uncommon in PAH and food consumption is adequate. Aim 2) Measure the stability over time in plasma carnitine levels in PAH patients. This aim will test the hypothesis that plasma carnitine is not affected by disease severity and is stable over time in PAH patients. The study will measure plasma carnitine concentration and markers of fatty acid oxidation at Visit 1 and Visit 2. 3) Perform a mechanistic pilot study using carnitine supplementation to enhance circulating carnitine in PAH. This small pilot study will test the hypothesis that carnitine supplementation increases plasma carnitine (primary endpoint) and will test for physiologic effects using six minute walk testing, echocardiography and plasma markers of lipid metabolism.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 or older.
* Diagnosed with idiopathic, heritable, simple congenital heart defect, or drug- or toxin-associated pulmonary arterial hypertension (PAH) according to World Health Organization consensus recommendations.
* Stable PAH-specific medication regimen for three months prior to enrollment. Subjects with only a single diuretic adjustment in the prior three months will be included. Adjustments in IV prostacyclin for side effect management are allowed.
* FEV1> or = 60% predicted and no more than mild abnormalities on lung imaging
* WHO Functional Class II-IV
* Ambulatory

Exclusion Criteria:

* Prohibited from normal activity due to wheelchair bound status, bed bound status, reliance on a cane/walker, activity-limiting angina, activity-limiting osteoarthritis, or other condition that limits activity
* Pregnancy
* Diagnosis of PAH etiology other than idiopathic, heritable, simple congenital heart defect, or associated with drugs or toxins
* Drug and toxin associated PAH patients with active drug use
* Prior diagnosis of cirrhosis
* Malignancy
* eGFR by MDRD <60mL/min
* Known allergy to l-carnitine supplements

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2021-09-29 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anna R Hemnes, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Yes
Since the data that will be produced involves patients with a disease process that is much in need of new treatment options and the investigators agree that data sharing is essential for expedited translation of research results into patient treatment options. A detailed data sharing plan is in place and available upon request. In brief:
  It is the investigator's plan to make data available at the time it is accepted for publication of the main findings from the final dataset through the use of a data enclave of our own design that would restrict our Data Analyst from sharing any information that would breach participant confidentiality. Potential researchers will contact the PI to discuss specific needs and how the data will be utilized. A formal approval process is in place to evaluate and complete such requests.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 2 years after study completion.
Access Criteria: * detailed written description of the project for which the data would be used
  * acknowledge in any publication resulting from the data, the source of the data, crediting the program support
  * agree to submit all papers or reports submitted for publication to the PI for review prior to submission

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Single arm study
Period: Overall Study
Arm/Group | Supplement
Started | 10
Visit 1 | 9
Completed | 8
Not Completed | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | Supplement
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.3 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 8
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 9
  More than one race | 0
  Unknown or Not Reported | 0
Functional Class [Count of Participants; unit: Participants] — The WHO functional classification for PAH has been modified from the well-known New York Heart Association functional classification. This functional classification is based on symptoms, with Class I being defined by no symptoms, Class II as having mild limitation in physical activity, Class III as having markedly limited physical activity and Class IV as being unable to perform any physical activity.
  Participants
    Functional Class I | 1
    Functional Class II | 8
    Functional Class III | 0
    Not evaluated | 1

OUTCOME MEASURES:

1. Primary Outcome: Plasma Carnitine Concentration
Description: Change in plasma Carnitine concentration from Visit 2 (Week 12) to Visit 4 (Week 14).
Time Frame: 2 weeks of intervention
Measure: Median (Inter-Quartile Range); unit: uM
Arm/Group | Supplement
Number analyzed (Participants) | 7
uM | 44 [37.3 to 48.7]

2. Secondary Outcome: Prevalence of Carnitine Supplement Use
Description: Quantify the prevalence of Carnitine supplement use of Carnitine in PAH patients by evaluating the number of study participants that report use of a daily carnitine supplement in baseline dietary reporting.
Time Frame: 12 weeks
Population: Number of participants reporting carnitine supplement use
Measure: Count of Participants; unit: Participants
Arm/Group | Supplement
Number analyzed (Participants) | 7
Participants
  Baseline | 0
  12 weeks | 0

3. Secondary Outcome: Carnitine Ingestion Use Through Food
Description: Measure oral ingestion of Carnitine in PAH patients by assessing food intake recorded by diary. Reports lacking meat, fish, and/or eggs are deemed "no ingestion by diet".
Time Frame: Reported week 1 (3 days leading up to visit 1) and week 12 (3 days leading up to visit 2).
Population: Number of subjects that ate a standard diet that included carnitine meat, fish and/or eggs, which provide Carnitine.
Measure: Count of Participants; unit: Participants
Arm/Group | Supplement
Number analyzed (Participants) | 7
Participants
  Week 1 | 7
  Week 12 | 7

4. Secondary Outcome: Six-minute Walk
Description: Mean change in meters walked pre- and post- carnitine on 6mwt
Time Frame: 14 weeks
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Supplement
Number analyzed (Participants) | 7
meters | 13.14286 (17.9)

5. Secondary Outcome: WHO Functional Class
Description: count of pre- and post-carnitine supplement and WHO functional class
Time Frame: 14 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Supplement
Number analyzed (Participants) | 7
Participants
  Pre-supplement: WHO functional class I | 3
  Pre-supplement: WHO functional class II | 4
  Post-supplement: WHO functional class I | 2
  Post-supplement: WHO functional class II | 5

6. Secondary Outcome: Patient Reported Side Effects
Description: Markers of tolerability of Carnitine supplement including presence of side effects, adverse events, and serious adverse events. Side effects to be reported beginning Visit 2, at carnitine start, and ended at Visit 4.
Time Frame: 2 weeks- between visit 2 and visit 4
Population: number of participants reporting side effects
Measure: Number; unit: participants
Arm/Group | Supplement
Number analyzed (Participants) | 7
participants | 1

7. Secondary Outcome: Echocardiography Measurements of TAPSE and RV Fractional Area
Description: Correlation of change in plasma Carnitine with change in markers of RV function including TAPSE and RV fractional area change
Time Frame: 14 weeks
Measure: Number (95% Confidence Interval); unit: correlation coefficient
Arm/Group | Supplement
Number analyzed (Participants) | 6
correlation coefficient
  TAPSE- Spearman | 0.543 [-0.480 to 0.940]
  RV fractional- Spearman | -0.086 [-0.839 to 0.780]
  TAPSE- Pearson | 0.736 [-0.187 to 0.969]
  RV fractional area- Pearson | 0.107 [-0.772 to 0.845]

8. Secondary Outcome: Stability of Plasma Carnitine
Description: Change in plasma carnitine from visit 1 to visit 2
Time Frame: 12 weeks- change from visit 1(week 1) to visit 2(week 12)
Measure: Median (Inter-Quartile Range); unit: uM change
Arm/Group | Supplement
Number analyzed (Participants) | 9
uM change | 2.708 [0.249 to 7.154]

ADVERSE EVENTS:
Time Frame: Participants were monitored for adverse events for a total of 16 weeks, from Visit 1 until 14 days following the last administration of study treatment.
Arm/Group | Supplement
All-Cause Mortality (participants affected / at risk) | 1/10
Serious Adverse Events (participants affected / at risk) | 1/10
Other Adverse Events (participants affected / at risk) | 3/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Supplement (N=10)
Chest pain (Cardiac disorders) | 1 (1) — Female with PMH significant for pulmonary hypertension who presents to the ED for chest pain.
Pericardial effusion (Cardiac disorders) | 1 (1) — During the participant's research visit echocardiogram, the technician identified a pericardial effusion (greater than that shown on ECHO in January).
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Supplement (N=10)
Foot fracture (Musculoskeletal and connective tissue disorders) | 1 (1) — Participant broke foot while on trial.
Respiratory symptoms (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Over-diuresed in setting of suspected viral illness
Cough, dyspnea with exertion, fatigue (General disorders) | 1 (1) — observation of increasing shortness of breath, chest tightness, fatigue, and cough following COVID booster vaccination

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-09-07): https://cdn.clinicaltrials.gov/large-docs/97/NCT04908397/Prot_SAP_001.pdf
  • Informed Consent Form (2022-04-19): https://cdn.clinicaltrials.gov/large-docs/97/NCT04908397/ICF_002.pdf